CLINICAL TRIAL: NCT06522659
Title: Evaluation of Clinical and Radiographic Outcomes of Surgically Treated Multiligamentous Knee Injuries
Acronym: MULTI-LIG
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: MULTI-LIG
Record Dates: First submitted 2024-07-11; First posted 2024-07-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Knee Ligament Injury; PCL - Posterior Cruciate Ligament Rupture; PROMs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiligament knee injuries are typically caused by high-energy mechanisms and are classified according to the number of ligaments involved using Schenk's classification (Knee Dislocation) into KD 1, KD 2, KD 3, and KD 4. These types of injuries can have devastating consequences on the individual's quality of life, affecting their ability to return to sports and perform daily activities.

In the literature, there is still no consensus on the management of these types of traumas, both due to the wide range of situations that can present to the orthopedic surgeon and the difficulty in their diagnostic and therapeutic framing. The main controversies concern the conservative or surgical management of the injuries and the timing of when to undertake surgical treatment, if at all.

The instability resulting from multiligament knee injuries is poorly tolerated by patients, who find their daily activities limited. It is also well known that this instability can dramatically accelerate the development of osteoarthritis, leading to the need for joint replacement surgery even in young individuals, thus increasing the likelihood of revisions and re-operations over time.

Due to the lack of standardized and satisfactory treatment, the economic cost of the outcomes of multiligament knee injuries is particularly high. A recent study by XXX showed that only XXX% of individuals are able to return to work. The rate of participation in sports is even lower, which has a long-term potential impact by increasing the risk of sedentary lifestyle-related diseases such as obesity, diabetes, and cardiovascular diseases.

The choice of surgical treatment aims to eliminate the patient's subjective feeling of instability and to repair, when possible, or reconstruct the injured ligament structures to reduce the risk of secondary osteoarthritis. Available studies in the literature are often case reports presenting short- and medium-term results of non-standardized surgical techniques with great heterogeneity in rehabilitation protocols, so the real long-term effectiveness of these treatments in terms of joint stability and osteoarthritis prevention is not known.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 65 years at the time of surgery
2. Male and female gender
3. Patients undergoing multiligamentous knee reconstruction from January 1, 2000, to December 31, 2019, at the Rizzoli Orthopedic Institute.

Exclusion Criteria:

1. Patients no longer reachable;
2. Patients who do not consent to be included in the study;
3. Pregnant women;
4. Presence of infection or hematologic, rheumatic, or coagulative disorders at the time of evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from all subjects treated surgically with multiligament knee reconstruction techniques from January 1, 2000, to December 31, 2019, at the Rizzoli Orthopedic Institute.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) | 5 years
  The IKDC form assesses knee function and symptoms across three domains: Symptoms (pain, stiffness, swelling, locking), Sports and daily activities, and Current knee function compared to before injury. It includes 10 questions: seven on symptoms, one on sports, one on daily activity difficulties, and one on current knee function. Scores range from 0 to 100, with higher scores indicating better knee function (excellent: 80-100, good: 60-80, fair: 30-60, poor: 0-30).

SECONDARY OUTCOMES:
Lysholm Knee Score | 5 years
  It is a validated measurement scale that assesses knee functionality through 8 items that determine the condition of the knee in response to the functional demands of daily life activities. This evaluation form is used to assess the surgical outcomes in patients who have undergone surgery for ligament or meniscal injuries of the knee.
  The final score is obtained by summing the various scores from the different items, ranging from 0 to 100. Scores are divided into subgroups: Excellent (95-100), Good (84-94), Fair (65-83), and Poor (<64).

OTHER OUTCOMES:
Visual Analog Scale (VAS) | 5 years
  It is a one-dimensional quantitative numerical scale for assessing pain on a 10-point scale. The scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at that specific moment. 0 means no pain, and 10 indicates the worst possible pain.
SF-36 (Short Form-36 Health Survey) | 5 years
  The SF-36 is the most well-known and widely used health-related quality of life measurement tool in international literature. It measures different health concepts through 36 multiple-choice questions. The data are aggregated into 8 scales that investigate: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Additionally, there is one question regarding changes in health status over the past year.
Tegner Score | 5 years
  The Tegner Score estimates the level of physical activity of an individual with a score ranging from 0 to 10, where 0 represents 'disability' and 10 represents 'participation in competitive sports, such as national or international level soccer.' This score is the most commonly used to define the activity level of patients with knee disorders. In the study, the Tegner Score will be completed directly by the investigator through an interview with the patient.
Time taken to return to work | 5 years
  The ability to return to work following the trauma will be assessed with a questionnaire, including the capacity to perform the same job duties.
Clinical evaluation | 5 years
  The stability of the operated knee will be globally assessed using routine knee evaluation tests.
Radiographic assessment | 5 years
  Clinical and imaging data will be collected from patients to assess osteoarthritis development and severity, along with any other radiographic abnormalities. If recent radiological records are not available as per study protocol in the last 12 months, a weight-bearing X-ray of the lower limbs (panoramic and lateral views of the operated knee) will be conducted. This aims to classify osteoarthritis severity using the Kellgren-Lawrence scale, which grades knee osteoarthritis from 0 (no visible changes) to 4 (severe joint space narrowing, bone sclerosis, and osteophyte formation).

CONTACTS AND LOCATIONS:
Locations (1):
- IRRCS Rizzoli Ortopedic Institute, Bologna, Italy